CLINICAL TRIAL: NCT03383913
Title: Use of Heart Rate Variability (HRV) Biofeedback for Symptom Management Among Sickle Cell Patients: Pilot Intervention
Brief Title: HRV-B for Symptom Management in Sickle Cell Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00066320
Record Dates: First submitted 2017-07-18; First posted 2017-12-27 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease
Keywords: Heart Rate Variability Biofeedback; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm baseline visit will include: Institutional Review Board (IRB) consent, PROMIS measure baseline and outcome assessments, instructions on placement of Firstbeat device and use of Firsbeat journal, resting HRV recording using Firsbeat software for 15 minutes, saliva collection, and distribution of actigraph watch to quantify sleep quality. Participants placed in the intervention arm will receive 4-6 weeks of Heart Rate Variability Biofeedback training. All measures will be repeated at the end of the six week period.
  Interventions: Behavioral: Heart Rate Variability Biofeedback
- Control (No Intervention): The control arm baseline visit will include: Institutional Review Board (IRB) consent, PROMIS measure assessments, instructions on placement of Firstbeat device and use of Firsbeat journal, resting HRV recording using Firstbeat software for 15 minutes, saliva collection, and distribution of actigraph watch to quantify sleep quality. The control group will receive their usual care for SCD and complete baseline and post-baseline outcome assessments without any HRV-B training. All measures will be repeated at the end of the six week period.

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback — Over a period of 4-6 weeks participants in the intervention arm will learn a series of breathing techniques to determine Heart Rate Variability's effects on physical function, anxiety, depression, fatigue, sleep disturbance, participation in social activities, pain interference and intensity.
  Arms: Intervention

SUMMARY:
This study will test the hypothesis that Heart Rate Variability Biofeedback (HRV-B) restores autonomic balance and reduces pain and other symptoms among patients with sickle cell disease (SCD).The specific aims of this study are to: (1) conduct a randomized, wait list controlled, pilot intervention trial to determine whether HRV-B increases HRV coherence among SCD participants (minimum N of 30, up to 50 total); (2) determine whether HRV-B reduces pain, stress, fatigue, depression or insomnia among SCD participants; and (3) determine whether increases in HRV coherence are associated improvements in pain, stress, fatigue, depression, or sleep among study participants.

DETAILED DESCRIPTION:
The purpose of this study is to see if Heart Rate Variability Biofeedback (HRV-B) can reduce chronic pain, stress, depression, anxiety, insomnia, loneliness, helplessness, physical limitations and pain medication dependence. HRV-B is an interactive procedure in which participants relax and breathe regularly while watching a computer screen. The computer screen provides feedback that helps people increase their heart rate variability, which is the difference from beat to beat. HRV-B is a complementary, non-pharmacologic therapy that is now being used to see if it can help sickle cell patients reduce their symptoms of pain, stress, insomnia, fatigue, or depression.

Participants will be randomly assigned to either an Intervention Group or a Comparison Group. Each group will have about 15-20 participants. The Intervention group will receive a baseline assessment including symptom questionnaires, up to six weekly HRV-B training sessions lasting about 45 minutes each, and a follow-up assessment including symptom questionnaires. There are 6-8 total visits for the intervention group and 2 for the control group. The Comparison Group will have a baseline assessment including symptom questionnaires, then six weeks with no training sessions, then a follow up assessment including symptom questionnaires. After the follow up assessment, the Comparison Group members will have the option of receiving the same treatment as the Intervention Group.

ELIGIBILITY:
Inclusion Criteria:

* SCD patients
* 10 years old
* English literate
* Patient recruited through Greenville Health System
* Any race or ethnicity
* Any sex

Exclusion Criteria:

* Conditions affecting HRV (paroxysmal supraventricular tachycardia, atrial fibrillation, myocardial infarction within 12 months, unstable angina)
* Medications that affect cardiac rhythm (angiotensin converting enzyme, calcium channel, or beta-adrenergic inhibitors)
* Pacemaker or defibrillator
* Heart transplant or by-pass surgery within 1 year
* Active seizure disorder or use of antiseizure/anticonvulsant medication specifically for seizures
* Dementia
* Moderate or severe head injury or stroke within 6 months
* Evidence of active substance abuse
* An uncontrolled major psychiatric disorder
* Cognitive disability that precludes participation
* Use of long acting (extended release) opioid medications; however, 'as needed' short acting opioid medication usage is allowable

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Measures | 4-6 weeks
  A comprehensive survey of physical function, anxiety, sleep disturbance, depression, fatigue, social roles, pain interference, and pain intensity are completed before the study begins and upon completion. Each domain is measured with a separate short form consisting of eight questions, with the exception of pain intensity, which is measured as a raw score of zero to ten. The scores of these surveys are combined. This number is then converted to a single PROMIS measure T score metric.

SECONDARY OUTCOMES:
Sleep Quality | 4-6 weeks
  Sleep quality will be quantified using wrist actigraph monitors that will be worn by the subject for seven days at the beginning and end of the study
C-Reactive Protein in saliva | 4-6 weeks
  Protein saliva samples will be collected by participants at baseline and at followup. Using an ELISA assay kit we will quantify inflammation mediators and C-Reactive Protein.

CONTACTS AND LOCATIONS:
Overall Officials: Aniket Saha, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Center for Integrative Oncology and Survivorship, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No